CLINICAL TRIAL: NCT05551546
Title: Effect of Functional Medicine Health Coaching on Self-Reported Measures of Physical and Emotional Health: A Randomized Controlled Trial.
Brief Title: Functional Medicine Health Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute for Functional Medicine (Other)
Collaborators: Functional Medicine Coaching Academy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EliminationDietRCT1
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Health Promotion
MeSH Terms: interventions — Elimination Diets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Medicine Health Coaching for Elimination Diet (Active Comparator): Participants randomized into the "Functional Medicine Health Coaching for Elimination Diet" arm will receive five remote health coaching sessions over 10 weeks in support of their progress through an elimination diet. All study arms will receive written elimination diet support materials.
  Interventions: Behavioral: Functional Medicine Health Coaching for Elimination Diet for Elimination Diet
- Self-guided Elimination Diet (Other): Participants randomized into the "Self-guided Elimination Diet" group will engage with the elimination diet without health coaching. All study arms will receive written elimination diet support materials.
  Interventions: Behavioral: Self-guided Elimination Diet

INTERVENTIONS:
Behavioral: Functional Medicine Health Coaching for Elimination Diet for Elimination Diet — All participants will receive 5 coaching sessions to support them through the elimination diet.
  First session: The foundation session is where the coach and participant begin to develop rapport and outline the participant's goals. This occurs before the start of the Elimination Diet for motivation, expectations, education, and preparation.
  Second session: This can occur during week 1 of the elimination diet to support working through the implementation.
  Third session: This session is recommended to occur during week 3 of the diet to prepare for the reintroduction of foods.
  Fourth session: A session is recommended while the participant is reintroducing foods as this is typically the most difficult part of the diet as participants may be experiencing symptoms to reactive foods.
  Fifth session: A wrap up session is recommended after all of the food re-introductions to support the participant with maintenance, goals to move forward, and reflection.
  Arms: Functional Medicine Health Coaching for Elimination Diet
Behavioral: Self-guided Elimination Diet — The Elimination Diet course materials include self-guided materials designed to guide participants through all phases of a comprehensive elimination diet, including preparation, elimination, and reintroduction phases.
  All participants in this wait-list control group will be presented via email with the opportunity to receive the five sessions of coaching (described above) at the conclusion of the study.
  Arms: Self-guided Elimination Diet

SUMMARY:
The goal of this research is to evaluate the feasibility and self-reported health outcomes of functional medicine health coaching in elimination diets among clinicians receiving training in functional medicine.

A randomized controlled clinical trial of a 5-session functional medicine coaching and elimination diet intervention will be conducted to achieve the purpose of this study. The research team hypothesizes that functional medicine health coaching to support the elimination diet will improve physical and mental health outcomes better than the control condition of a self-guided elimination diet.

ELIGIBILITY:
Inclusion Criteria:

* Agree to adopt the elimination diet as outlined by study sponsor with no pre-planned interruption
* Able to understand and write English
* Voluntarily consent to the study and understand its nature and purpose including potential risks and side effects

Exclusion Criteria:

* Eating disorders within the past 10 years
* Currently pregnant or breastfeeding
* Nursing home residents, other institutionalized persons, prisoners, any other vulnerable participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline PROMIS-Global Health score | Change from baseline at 10 weeks
  The PROMIS Global Health is a 10-item survey (PROMIS-10) is measure of health status that spans physical, mental, and social domains from the patient perspective, allowing clinicians and researchers to capture the complex and heterogeneous nature of the populations.

SECONDARY OUTCOMES:
Change from baseline Medical Symptoms Questionnaire (MSQ) score | Change from baseline at 10 weeks
  The Medical Symptoms Questionnaire is a multi-system inventory that rates symptom severity on a 0-4 scale. The MSQ has been used to track subjective responses of patients to treatment in both clinical and research settings.
Adherence/compliance to the elimination diet | At 10 weeks
  The Adherence/compliance assessment is a 0-10 scale that asks the participant one question to self-rate how well they followed the Elimination Diet. This has been used in the Healthy Diet and Lifestyle Study pilot, a randomized trial.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Scheinbaum, PhD, Principal Investigator — Functional Medicine Coaching Academy
Locations (1):
- The Institute for Functional Medicine, Federal Way, Washington, United States

IPD SHARING:
Plan to Share IPD: No